CLINICAL TRIAL: NCT05238818
Title: Single Arm Phase I Trail of Autologous Tumor Infiltrating Lymphocyte Injection (GT202) in the Treatment of Metastatic or Recurrent Gynecological Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: XinWu (Other)
Responsible Party: Sponsor-Investigator, XinWu, Department Director, Obstetrics & Gynecology Hospital of Fudan University
Organization: Obstetrics & Gynecology Hospital of Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUOBGY2021-196
Record Dates: First submitted 2022-02-09; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Metastatic or Recurrent Gynecological Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT202 in Metastatic or Recurrent Gynecological Tumor patients (Experimental): Autologous Tumor Infiltrating Lymphocyte Injection (GT202) will be infused at 1.0×10^8 cells, 5.0×10^8 cells and 2.0×10^9 cells in metastatic or recurrent gynecological tumor patients.
  Interventions: Biological: Autologous Tumor Infiltrating Lymphocyte Injection (GT202)

INTERVENTIONS:
Biological: Autologous Tumor Infiltrating Lymphocyte Injection (GT202) — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. T cells then are manufactured to express mbIL-12. After lymphodepletion, patients are infused with GT202 followed by IL-2.

SUMMARY:
A prospective, open-label, non-randomized, Phase 1 study evaluating autologous tumor infiltrating lymphocyte injection (GT202) in the treatment of metastatic or recurrent Gynecological tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary participation and sign informed consent
* 2.Must be ≥ 18 and ≤70 years at the time of consent
* 3.Must be diagnosis of unresectable Metastatic or Recurrent Gynecological Tumors (limited to cervical cancer, ovarian cancer and endometrial cancer)
* 4.Must have progressed following at least one line of standard treatment, and there is no alternative effective treatment or alternative effective treatment plan rejected by patient (effective treatment refers to the latest version of diagnosis and treatment guidelines for various cancers)
* 5.At least one resectable lesion (or invaded superficial lymph nodes, or aggregate of lesions resected) of a minimum 0.5cm3 for resection to generate TIL. Minimally invasive surgery is preferred. This lesion cannot be in previously irradiated areas or other local therapy.
* 6.At least one another measurable target lesion after resection, as defined by RECIST v1.1. Lesions in previously irradiated areas (or other local therapy) should not be selected as target lesions, unless treatment was ≥ 3 months prior to screening, and there has been demonstrated disease progression in that particular lesion.
* 7.ECOG=0 or 1
* 8.Estimated life expectancy of ≥ 12 weeks
* 9.Patients must have adequate organ function:

  1. hematologic parameters: Absolute neutrophil count (ANC) ≥ 1.5×109/L Lymphocyte counts（LC）>0.5×109/L Platelet ≥100×109/L Hemoglobin (Hb) ≥ 90g/L
  2. AST, ALT and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN), TBIL (total bilirubin)≤1.5×ULN, except following:

patients with liver metastasis: AST, ALT≤ 5 times ULN; Patients with liver metastasis or bone metastasis: alkaline phosphatase≤5 times ULN; Patients with Gilbert syndrome: TBIL≤3.0 mg/dL; Estimated creatinine clearance (eCrCl) ≥ 45 mL/min using the Cockcroft-Gault formula, or serum creatinine in normal range; d) APTT≤1.5×ULN, while INR or PT≤1.5×ULN; e) LVEF ≥50%; f) FEV1≥60%;

* 10.Patients of childbearing potential or their partners of childbearing potential must be willing to take the appropriate precaution to avoid pregnancy or fathering a child for the duration of the study and practice an approved, highly effective method of birth control during treatment and for 12 months after receiving the last protocol-related therapy. Non surgically sterilized female subjects of reproductive age must be negative for serum hCG testing within 7 days prior to cell infusion;
* 11.Patients must have recovered from all prior therapy-related adverse events (AEs) to ≤ Grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] v5.0), except for alopecia or vitiligo, prior to enrollment (tumor resection). Patients with documented ≥ Grade 2 diarrhea or colitis as a result of previous treatment with immune checkpoint inhibitor(s) must have been asymptomatic for at least 6 months and/or had a normal colonoscopy post-immune checkpoint inhibitor treatment, by visual assessment, prior to tumor resection;
* 12.Before resection, the imaging evidence of disease progress after prior line treatment should be documented.

Exclusion Criteria:

* 1. Patients with symptomatic and/or untreated CNS metastases (Patients with definitively treated brain metastases may be considered for enrollment and must be stable for ≥ 14 days without drug treatment and steroid-dependent) ;
* 2. Failure of surgery and / or radiotherapy to relieve spinal cord compression;
* 3. Uncontrolled tumor related pain judged by the investigator. Subjects requiring pain medication must have had a stable pain medication regimen at the time of enrollment; symptomatic lesions amenable to palliative radiotherapy should have completed treatment before enrollment;
* 4. Interstitial pneumonia or clinically significant active pneumonia, or other respiratory disease severely affecting lung function;
* 5. Any active autoimmune disease; a history of autoimmune disease or disease requiring treatment with systemic steroids or immunosuppressive drugs;
* 6. Patients with a history of significant cardiovascular disease, including: 1) Congestive heart failure (NYHA functional classification > Class 2); 2) Unstable angina; 3) myocardial infarction occurred in past 3 months; 4) Any supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
* 7. Arterial/venous thrombotic events within 5 months prior to enrollment, such as: cerebrovascular accident, deep vein thrombosis and pulmonary embolism occurring;
* 8. Patients with active tuberculosis infection within 1 year before enrollment, or with a history of active tuberculosis infection beyond 1 year before but without standard treatment;
* 9. Active infections requiring treatment with systemic anti-infectives (except for topical antibiotics); or those with unexplained fever > 38.5℃ occurring during the screening period, except for tumor fever;
* 10. Patients with a history of immunodeficiency, including HIV seropositivity;
* 11. Patients with active hepatitis B or C. Patients with seropositive HBsAg or HBcAb can be enrolled while negative HBV DNA. Patients with seropositive HCV antibody can be enrolled while negative HCV RNA. If potential carriers enrolled, proper anti-virus treatment and regular nucleotide test should be arranged.
* 12. Patients with intractable or intractable epilepsy, ascites beyond drug control, portal vein tumor thrombus, gastrointestinal bleeding caused by gastric fundus or esophageal varices, increased risk of bleeding caused by portal hypertension, and active gastrointestinal bleeding
* 13. Patients who have received an organ allograft or prior cell transfer therapy;
* 14. Patients who have a history of hypersensitivity to any component or excipient of GT202 or other study drugs: autologous tumor infiltrating lymphocytes, cyclophosphamide, fludarabine, IL-2, dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40 and antibiotics (beta lactam antibiotics, gentamicin);
* 15. Known psychiatric disorders, alcohol, drug or substance abuse;
* 16. Any disease or condition (any other condition, metabolic disorder, physical exam result, or abnormal laboratory test result) that could lead to reasonable doubt that would prohibit the use of a trial drug, or affect the interpretation of study results, or put the patient at high-risk treatment;
* 17. Patients who are pregnant or breastfeeding;
* 18. Other circumstances that investigator assessed could affect the safety of subjects.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Types and incidence of Dose-limiting toxicity (DLT) | up to 28 days after GT202 infusion
  Dose-limiting toxicity (DLT) will be collected and graded according to CTCAE v5.0
Types and incidence of adverse events (AEs) ，serious adverse events (SAEs) and adverse events of special interest (AESI) | Up to 2 years after GT202 infusion
  AE will be collected and graded according to CTCAE v5.0
Maximum tolerated dose | up to 28 days after GT202 infusion
  Evaluate the Maximum tolerated dose of GT202 in Metastatic or Recurrent Gynecological Tumors patients

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 6 weeks, 12 weeks, 18 weeks, 24 weeks after GT202 infusion
  ORR will be calculated as the percentage of patients who achieved partial response (PR) or better.
Duration of Response (DOR) | Up to 2 years after GT202 infusion
  Time from first response to disease progression or death from any cause
Progression-free Survival (PFS) | Up to 2 years after GT202 infusion
  PFS will be calculated as the time from GT202 infusion to disease progression or death from any cause (whichever occurs first).
Overall Survival (OS) | Up to 2 years after GT202 infusion
  Time from GT202 infusion to time of death due to any cause
Disease Control Rate (DCR) | up to 6 weeks, 12 weeks, 18 weeks, 24 weeks after GT202 infusion
  DCR will be calculated as the percentage of patients who achieved Stable Disease(SD) or better.

CONTACTS AND LOCATIONS:
Overall Officials: xin wu, PHD, Principal Investigator — The Obstetrics and Gynecology Hospital of Fudan University
Locations (1):
- The Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No